CLINICAL TRIAL: NCT04648930
Title: Special Drug Use Observational Study of Xolair in Patients With Severe to Most Severe Seasonal Allergic Rhinitis Aged ≥ 12 Years and < 18 Years Whose Symptoms Were Inadequately Controlled Despite to Conventional Therapies
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025F1401
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Allergic Rhinitis
Keywords: Xolair; seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xolair: S.C. Injection
  Interventions: Drug: Xolair

INTERVENTIONS:
Drug: Xolair — There was no treatment allocation. Patients administered Xolair by prescription that started before inclusion of the patient into the study were enrolled.
  Other Names: Omalizumab

SUMMARY:
This was a multicenter, uncontrolled, open-label, special drug use study to investigate the safety and efficacy of Xolair by collecting data in its clinical setting in patients with severe to most severe seasonal allergic rhinitis aged ≥ 12 years and < 18 years whose symptoms were inadequately controlled despite to conventional therapies and used Xolair.

DETAILED DESCRIPTION:
The observation period lasted for up to 24 weeks, with Day 1 defined as the start date of Xolair treatment. It should be noted that, because the duration of Xolair treatment depends on the pollen dispersal situation and other factors, patients who completed or discontinued Xolair treatment before the visit at 24 weeks after the start of treatment were followed up until the date of last dose of Xolair + 30 days, and the results were recorded in the CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who used Xolair in accordance with the instructions of package insert
2. Patients aged ≥ 12 years and < 18 years at the start of Xolair
3. Patients who used Xolair for the following indication:

Indication: seasonal allergic rhinitis (only patients with severe to most severe symptoms whose symptoms were inadequately controlled despite to conventional therapies) 4. Patients having provided written consent to participate in this study before the start of Xolair in the relevant pollen season, in person and from their legally acceptable representative (legal representative)

Exclusion Criteria:

1. Patients with a history of hypersensitivity to any of the Xolair ingredients

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population was patients with seasonal allergic rhinitis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Proportions of patients with Adverse events (AEs), Serious AEs, AEs leading to discontinuation of Xolair treatment, Adverse drug reactions (ADRs), Serious ADRs, ADRs leading to discontinuation of Xolair treatment | up to 24 weeks
  The number of patients with each events and incidences (%) will be calculated by System Organ Class (SOC) and Preferred Term (PT).
  SAEs are defined as AEs meeting the criteria of seriousness and adverse events with a fatal outcome.
  ADRs are defined as AEs for which a causal relationship with Xolair is not ruled out by the investigator.

SECONDARY OUTCOMES:
Overall improvement rate of disease by physicians | week 24
  The investigator comprehensively assessed the therapeutic effect of Xolair on seasonal allergic rhinitis at the last visit on the basis of the patient's condition before the start of Xolair and during the clinical course thereafter, as "markedly improved", "moderately improved", "slightly improved", "no change" or "worsened"
Disease severity of seasonal allergic rhinitis | Up to 24 weeks
  The investigator comprehensively assessed the severity of seasonal allergic rhinitis on the basis of each seasonal allergic rhinitis symptom, test results, and the degree of visually examined local changes at each visit, as "very severe", "severe", "moderate", "mild" or "no symptom"
Individual symptom severity of seasonal allergic rhinitis | Up to 24 weeks
  The investigator assessed the severity of each seasonal allergic rhinitis symptom(sneezing, nasal discharge, nasal obstruction, difficulty in daily activity) at each visit in accordance with the criteria in the Practical Guideline for the Management of Allergic Rhinitis in Japan (2016)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Japan (13):
  - Novartis Investigative Site, Inazawa, Aichi-ken
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Inzai, Chiba
  - Novartis Investigative Site, Chikusei, Ibaraki
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Neyagawa, Osaka
  - Novartis Investigative Site, Chiyoda City, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Nagasaki
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Saitama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CIGE025F1401 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18085